CLINICAL TRIAL: NCT06659809
Title: 2-Brain Regulation to Achieve Improved Neuroprotection During Early Development (2- BRAINED)
Brief Title: 2-Brain Regulation to Achieve Improved Neuroprotection During Early Development
Acronym: 2-BRAINED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS National Neurological Institute "C. Mondino" Foundation (Other)
Collaborators: IRCCS Eugenio Medea (Other); National Research Council, Institute of Clinical Physiology, Italy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2-BRAINED
Record Dates: First submitted 2024-05-29; First posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-05

CONDITIONS: Premature Birth
Keywords: preterm birth; EEG; hyperscanning; video-feedback; early intervention; brain-to-brain co-regulation
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- VPT infants and their caregivers randomly allocated to the intervention arm (VPT-VF) (Experimental): Mother-infant dyads will partecipate in 6 weekly 1-hour sessions of Tele-care video-feedback intervention
  Interventions: Behavioral: Tele-care video-feedback intervention (TVFI)
- VPT infants and their caregivers randomly allocated to the care as usual arm (VPT-CU) (No Intervention): Usual care; no VF intervention. This arm will act as a control group matched to preterm conditions of VPT-VF.
- FT infants and their caregivers (FT-CG) (No Intervention): Usual care; no VF intervention. This arm will act as an additional control group unmatched to preterm conditions.

INTERVENTIONS:
Behavioral: Tele-care video-feedback intervention (TVFI) — The TVFI 6 weekly sessions are organized in two subsequent phases: 4 sharing the focus sessions and 2 integration sessions. Sharing the focus sessions are dedicated to the discussion between the psychologist and the mother of specific themes related to parenting and parent-infant interaction: physical stimulation, responsiveness, teaching, and parenting experience. The goal of the sharing the focus sessions is to develop insights about the infants' behavioral signals, the best ways to provide stimulations and get in touch, strategies to promote emotion regulation, and to sustain cognitive and behavioral achievements. In the subsequent two integration sessions, the mother plays with the infant while the psychologist provides guidance based on topics previously discussed during the first four sessions. The goal is to promote a pragmatical translation of the insights developed during the sharing the focus sessions into the interactive exchanges between the mother and the infant.
  Arms: VPT infants and their caregivers randomly allocated to the intervention arm (VPT-VF)

SUMMARY:
Each year 15 million infants are born preterm (PT). Even without severe comorbidities, they are exposed to sensory stress during the Neonatal Intensive Care Unit (NICU) stay and are at greater risk of neurodevelopmental problems compared to full-term (FT) counterparts in the short- and long-term period. Altered biobehavioral interpersonal synchrony patterns are documented in PT parent-infant dyads and might contribute to detrimental outcomes. Electroencephalographic (EEG) hyperscanning provides innovative real-time central biomarkers of brain-to-brain co-regulation; it was never applied to PT mother-infant dyads. Early parenting video-feedback (VF) interventions promote at-risk infants' neurodevelopment, yet action mechanisms are partially unknown. The present longitudinal project aims (a) to compare indexes of brain-to-brain co-regulation between dyads of full-term (FT) and VPT infants interacting with their mothers and (b) to investigate the effect of an early post-discharge VF intervention on the brain-to-brain co-regulation indexes of VPT dyads. This study will establish translational hyperscanning as a new field of innovative research with crucial clinical implications.

DETAILED DESCRIPTION:
Very preterm (VPT) birth is a major risk condition for child neurological and behavioral development and as well as for parental well-being, mainly due to multiple sources of stress (e.g., separation and pain exposure) during the hospitalization. Even in absence of severe critical medical comorbidities, VPT infants and their parents are exposed to multiple stress sources during the stay in the hospitalization in the Neonatal Intensive Care Unit (NICU), including early parent-infant separation and pain. Early parenting video-feedback (VF) interventions focused on promoting parent-infant closeness through the video-feedback (VF) approach methodology have proven effective in promoting child development and parental well-being. Electroencephalography (EEG) hyperscanning paradigms allow the assessment of brain-to-brain co-regulation during live interaction between infants and parents and hold promises to highlight mechanisms behind the interactive benefits of early VF parenting interventions. The 2-Brain Regulation to Achieve Improved Neuroprotection during Early Development (2-BRAINED) research project aims (a) to compare indexes of brain-to-brain co-regulation between dyads of full-term (FT) and VPT infants interacting with their mothers and (b) to investigate the effect of an early post-discharge VF intervention on the brain-to-brain co-regulation indexes of VPT dyads.

The 2-BRAINED project is a randomized-controlled trial (RCT) with three arms (see arm description). VPT (gestational age below 35 weeks) and FT (gestational age above 37 weeks) dyads will be enrolled at birth and the former will be randomly allocated to one of two arms: VF intervention or care as usual. The VF intervention will be delivered during the first three months after NICU discharge, consisting of and consists of 8 weekly remote VF sessions focused on sensory, behavioral, cognitive, and affective dimensions of parenting. Before and after the intervention, videotaped mother-infant interaction will provide pre-post behavioral data to assess the short-term effectiveness of the VF intervention. Videos will be micro-analytically coded for infant's and caregivers' target behaviors.

Mothers of VPT and FT infants will fill in questionnaires focused on maternal well-being (symptoms of depression [Beck Depression Inventory, BDI; Beck et al.,1961] and anxiety [State-Trait Anxiety Inventory, STAI-Y, Spielberg, 1983]), parenting (parental stress and mother-infant bonding [Parenting Stress Index, PSI; Abidin, 1983]), and infant development (language [Italian adaptation of the MacArthur-Bates Communicative Development Inventory; Caselli & Casadio, 1995]; temperament [Infant Behavior Questionnaire Revised, IBQ-R, Gartstein et al., 2003] and sensory profile [Sensory Profile 2, SP-2, Dunn, 2014]) at 3, 6 and 9 months (corrected age, CA).

At 9 months CA, all dyads will take part in a lab-based 5-min EEG- hyperscanning Still-Face task (Tronick et al., 1978; Provenzi et al., 2016) in the laboratory to assess brain-to-brain co-regulation, during which EEG activity from both the interactive partners will be recorded using two 32-electrode caps linked with two PC-connected wireless amplifiers (Smarting mBrainTrain) that will assure complete freedom of movements. Several indexes used to measure of brain-to-brain co-regulation will be tested and compared, including Phase-Locking Value (PLV), Amplitude-Amplitude Coupling (AAC) and imaginary coherence (ICoh). These indexes will be used to compare brain-to-brain co-regulation indexes (a) between PT and FT infants to test difference in interpersonal neurophysiological attunement in typical and at-risk infants as well as (b) between PTCU and PTVF. Moreover, best-fitting synchrony indexes will be used in a path analysis model testing the mediating role of brain-to-brain co-regulation indexes on the effects of VF early parental intervention on the short- and long-term outcomes. A prediction model will be implemented to predict outcomes on the basis of both clinical and EEG measures.

ELIGIBILITY:
Inclusion Criteria:

* infants' (corrected) age between birth and 3 months;
* parental age greater than 18 years;
* parental mastery of Italian language;
* parents living together with the infant;

Exclusion Criteria:

* infant's major comorbidities (e.g., genetic syndromes, malformations, brain injuries);
* parental psychiatric diagnoses;

Max Age: 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 159 (Estimated)
Dates: Start 2023-04-24 (Actual); Primary Completion 2025-12-24 (Estimated); Study Completion 2026-04-24 (Estimated)

PRIMARY OUTCOMES:
Phase-Locking Value (PLV) | 9 months (infant's corrected age)
  EEG index of brain-to-brain co-regulation among PT and FT parent-infant dyads
Amplitude-Amplitude Coupling (AAC) | 9 months (infant's corrected age)
  EEG index of brain-to-brain co-regulation among PT and FT parent-infant dyads
Imaginary Coherence (ICoh) | 9 months (infant's corrected age)
  EEG index of brain-to-brain co-regulation among PT and FT parent-infant dyads

SECONDARY OUTCOMES:
Parental NICU-related stress | NICU discharge T1 (only VPT)
  Parental Stressor Scale - NICU (PSS-NICU) (Miles, 1993).
Sensory profile | 3 months (infant's corrected age) T2
  Sensory Profile-2 (SP-2) (Dunn, 2014)
Sensory profile | 6 months (infant's corrected age) T3
  Sensory Profile-2 (SP-2) (Dunn, 2014)
Sensory profile | 9 months (infant's corrected age) T4
  Sensory Profile-2 (SP-2) (Dunn, 2014)
Anxiety symptoms | 3 months (infant's corrected age) T2
  State-Trait Anxiety Inventory (STAI-Y) (Spielberger et al., 1983)
Anxiety symptoms | 9 months (infant's corrected age) T4
  State-Trait Anxiety Inventory (STAI-Y) (Spielberger et al., 1983)
Depression symptoms | 3 months (infant's corrected age) T2
  Beck Depression Inventory (BDI-II) (Beck et al., 1996)
Depression symptoms | 9 months (infant's corrected age) T4
  Beck Depression Inventory (BDI-II) (Beck et al., 1996)
Parenting stress | 3 months (infant's corrected age) T2
  Parenting Stress Index - Short Form (PSI-SF) (Abidin, 1995)
Parenting stress | 6 months (infant's corrected age) T3
  Parenting Stress Index - Short Form (PSI-SF) (Abidin, 1995)
Parenting stress | 9 months (infant's corrected age) T4
  Parenting Stress Index - Short Form (PSI-SF) (Abidin, 1995)
Temperament | 3 months (infant's corrected age) T2
  Infant Behavior Questionnaire-Revised (IBQ-R) very short form (Gartstein & Rothbart, 2003)
Temperament | 6 months (infant's corrected age) T3
  Infant Behavior Questionnaire-Revised (IBQ-R) very short form (Gartstein & Rothbart, 2003)
Temperament | 9 months (infant's corrected age) T4
  Infant Behavior Questionnaire-Revised (IBQ-R) very short form (Gartstein & Rothbart, 2003)
Language and communication development | 3 months (infant's corrected age) T2
  Italian adaptation of the MacArthur-Bates Communicative Development Inventory (MB-CDI Fenson et al., 2007)
Language and communication development | 6 months (infant's corrected age) T3
  Italian adaptation of the MacArthur-Bates Communicative Development Inventory (MB-CDI Fenson et al., 2007)
Language and communication development | 9 months (infant's corrected age) T4
  Italian adaptation of the MacArthur-Bates Communicative Development Inventory (MB-CDI Fenson et al., 2007)

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Scientific Institute IRCCS E. Medea, Bosisio Parini
  - CNR Pisa, Pisa

IPD SHARING:
Plan to Share IPD: Yes
Raw data will be made available upon request through Zenodo repository
Supporting Information: SAP
Time Frame: After study completion
Access Criteria: Researchers will be able to access the raw data and the supporting information through the Zenodo repository upon request and after sharing an analysis plan